CLINICAL TRIAL: NCT05751395
Title: Siting Central Venous Catheters Precisely by Means of the ECG Method - A Study to Prove Reliability -
Brief Title: Siting Central Venous Catheters Precisely While Performing the Access Procedure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Deutsche Interdisziplinäre Vereinigung für Intensiv- und Notfallmedizin (Other)
Responsible Party: Principal Investigator, Wolfram Schummer, MD, PhD, Principle Investigator, Deutsche Interdisziplinäre Vereinigung für Intensiv- und Notfallmedizin
Other Study IDs: U1111-1285-5359
Record Dates: First submitted 2022-12-06; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Central Venous Catheter
Keywords: Central venous catheter; Double cannulation; ECG method (intravascular ECG); CVC tips; Verification technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill Patients in severe Multiple Organ Dysfunction: Critically ill Patients in severe Multiple Organ Dysfunction in need of a second Central Venous Catheter (CVC) for e.g. blood purification techniques
  Interventions: Device: Central Venous Access

INTERVENTIONS:
Device: Central Venous Access — Critically ill patients in severe MODS need a CVC and in some cases also a second line for e-g- blood purification techniques.
  All CVCs are positioned via the ECG method with the CVC tip placed at P-max. Within 24 h a chest radiograph is obtained for assessment of the CVCs, especially their tips.

SUMMARY:
For central venous catheters (CVC) to function properly, optimal tip location is of utmost importance.

One technique to verify CVC position is the ECG method. Nowadays, the ECG method is applied using the maximum P-wave amplitude (P-max).

The hypothesis is that a method believed to be precise in assessing CVC position can provide the same results for CVC tip positions regardless of their respective insertion sites.

Can the ECG method (at P-max) provide the same results for the position of CVC tips regardless of their insertion site?

DETAILED DESCRIPTION:
Only critically ill patients with multiple organ dysfunction are eligible for the study. Another condition is a prerequisite for reliable illustration of the results, i.e. at least two central venous lines has to be in place. All catheters are to be placed using the ECG method with the CVC tip at P-max. In all patients, a chest X-ray has to be performed within 24 hours of line insertion to assess the CVC positions.

The University's Institutional Review Board (IRB) registered and approved the study protocol (1518-03/05). The requirement for written informed consent was waived by the IRB.

Central venous catheters (CVC) play an important role in the management of critically ill patients by allowing measurement of haemodynamic variables that cannot be measured accurately by non-invasive means and by allowing delivery of medications and nutritional support that cannot be given safely through peripheral venous catheters. Unfortunately, these catheters are not without potential for harm. The insertion procedure in particular carries the risk of serious mechanical complications, though ultrasound imaging may dramatically reduce this risk.

For the catheter to function properly, tip location is of utmost importance. Inserting the tip too far into the right atrium raises serious risks of arrhythmias or even pericardial tamponade. Inserting it too shallowly - in the innominate vein or the upper third of the superior vena cava - poses the risk of intimal damage and consequently venous thrombosis, fibrin sleeve formation, and persistent withdrawal occlusion. Even with correct initial positioning, these catheters are prone to tip migration. However, the risk of erosion and even perforation of the vein wall also should not, in the light of their intensity, be ignored.

The ECG method of siting CVC tips has undergone marked development over recent decades. At present, the ECG method with its new interpretation - CVC tip at the maximum P-wave amplitude (P-max) - is a stable and reliable bedside method for positioning CVC tips exactly at the transition of the right atrium (RA) and superior vena cava (SVC) in patients in sinus rhythm. This is the only method that directly enables the operator to assess the correct CVC position during insertion. This study investigates the hypothesis that a method believed to be a precise approach to assessing CVC position can provide the same results for the position of two CVC tips regardless of respective insertion sites.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients in severe multiple organ dysfunction in need for a second CVC (e.g. for blood purification technique)

Exclusion Criteria:

* Patient selection not fulfilled a/o no need for a second CVC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only critically ill patients with multiple organ dysfunction treated in an ICU are eligible for the study. Another condition is a prerequisite for reliable illustration of the results, i.e. at least two central venous lines has to be in place. This implies that only patients in need of a second CVC (eg. for blood purification techniques) can be included into the study. All catheters are to be placed using the ECG method with the CVC tip at P-max. In all patients, a chest X-ray has to be performed within 24 hours of line insertion to assess the CVC positions.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
CVC tips are expected to be at the same level +/- 5 mm | Day 1
  CVCs placed by means of ECG method at P-max

SECONDARY OUTCOMES:
Difference between the level of CVC tips (expected to be at one level +/- 5mm) depending on chosen access site combination (e.g. right internal jugular vein versus left subclavian vein) | Day 1
  CVCs placed by means of ECG method at P-max

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Schummer, MD, PhD, Principal Investigator — Friedrich Schiller University
Locations (2):
- Germany (2):
  - Helios-Spital, Überlingen, Baden-Wurttemberg
  - University Clinic Leipzig, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: No
age gender height weight BMI CVC tip difference Access site and side

REFERENCES:
- [Result] Kremser J, Kleemann F, Reinhart K, Schummer W. Optimized method for correct left-sided central venous catheter placement under electrocardiographic guidance. Br J Anaesth. 2011 Oct;107(4):567-72. doi: 10.1093/bja/aer189. Epub 2011 Jun 22. PMID 21697183
- [Result] Wirsing M, Schummer C, Neumann R, Steenbeck J, Schmidt P, Schummer W. Is traditional reading of the bedside chest radiograph appropriate to detect intraatrial central venous catheter position? Chest. 2008 Sep;134(3):527-533. doi: 10.1378/chest.07-2687. Epub 2008 Jul 18. PMID 18641117
- [Result] Schummer W, Schummer C, Schelenz C, Schmidt P, Frober R, Huttemann E. [Modified ECG-guidance for optimal central venous catheter tip positioning. A transesophageal echocardiography controlled study]. Anaesthesist. 2005 Oct;54(10):983-90. doi: 10.1007/s00101-005-0886-2. German. PMID 16003543